CLINICAL TRIAL: NCT04737434
Title: The Effect of Extremely Low Frequency Electromagnetic Field Device Improving Sleep Quality and Stress
Brief Title: The Effect of Extremely Low Frequency Electromagnetic Field Device Improving Sleep and Stress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Tsai-Wei Huang, Associate Professor, Taipei Medical University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: N202006078
Record Dates: First submitted 2021-01-07; First posted 2021-02-03 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Stress; Sleep Quality; Fatigue; Extremely Low Frequency Electromagnetic Field Device; Schumann Resonance
Keywords: extremely low frequency electromagnetic field device; Stress; sleep quality; fatigue; HRV; Low Energy Emission Therapy; Schumann Resonance
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extremely low frequency electromagnetic field device (Experimental): with extremely low frequency electromagnetic wave
  Interventions: Device: Extremely low frequency electromagnetic field device
- electromagnetic field with no wave (Placebo Comparator): electromagnetic field with no wave
  Interventions: Device: electromagnetic field with no wave

INTERVENTIONS:
Device: Extremely low frequency electromagnetic field device — with extremely low frequency electromagnetic wave deliver or not to participants during sleep.
  Arms: Extremely low frequency electromagnetic field device
Device: electromagnetic field with no wave — electromagnetic field with no wave
  Arms: electromagnetic field with no wave

SUMMARY:
The purpose of this study is to explore the effects of extremely low frequency electromagnetic waves on improving stress and sleep quality. Experimental studies, pre- and post-test double-blind crossover tests are adopted. The selected subjects include: patients in the sleep center of the Taipei Medical University Hospital and the Department of Nursing and Bachelor of Taipei Medical University There are about 100 students in the post-nursing department. They are randomly assigned to groups A and B using a computer. The experiment period is two weeks. The two groups will take a pre-questionnaire test in the afternoon of the first day of the experiment and wear wearable bracelets. Group A first After getting the device with low-frequency electromagnetic field, group B first got the device without low-frequency electromagnetic field. The appearance of the two is the same. The bracelet is worn from the afternoon of the first day to the afternoon of the fourth day, a total of three days, and the device is withdrawn at the end of the first stage The two groups exchanged, repeat the steps to complete the second stage, after the end of the post-test, the two groups plug in the device half an hour before going to bed every day, and put it on the bedside table about 20cm away from the head, and then turn off the device after getting up. The research tools are basic attribute questionnaires, sleep quality scales, sleep diaries, smart care VIP bracelets, and EEG. Among them, the wearable bracelet can monitor the stress index, fatigue index, calories burned, and walking steps. Then SPSS 22.0 software is used for data file building and statistical analysis. The data is analyzed by descriptive statistics and inferential statistics. The expected result is that the experimental group and the control group have significant differences in reducing stress and improving sleep quality, which can relieve stress and improve sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* under 20 years old,great mental health,BMI is between 18.5~24(normal range).

Exclusion Criteria:

* Cognitive disturbance, confusion, pregnancy, alcohol and caffeine addiction.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-31 (Actual); Primary Completion 2023-01-25 (Estimated); Study Completion 2023-01-25 (Estimated)

PRIMARY OUTCOMES:
sleep quality | Baseline
  Questionnaire with PSQI(Pittsburgh Sleep Quality Index)
sleep quality | 2 weeks
  Questionnaire with PSQI(Pittsburgh Sleep Quality Index)

SECONDARY OUTCOMES:
stress level | Baseline
  Questionnaire with Perceived Stress Scale
stress level | 2 weeks
  Questionnaire with Perceived Stress Scale
fatigue levels | Baseline
  Questionnaire with VAS(Visual analogue scale) for fatigue level
fatigue levels | 2 weeks
  Questionnaire with VAS(Visual analogue scale) for fatigue level
HRV(Heart rate variability) level | Baseline
  Device measure including heart rate variability index, heart rate, etc.
HRV(Heart rate variability) level | 2 weeks
  Device measure including heart rate variability index, heart rate, etc.
EEG (Electroencephalography) power | Baseline
  a small portable EEG Device measure record including α, β, θ, δ wave and change style and time.
EEG (Electroencephalography) power | 2 weeks
  a small portable EEG Device measure record including α, β, θ, δ wave and change style and time.

CONTACTS AND LOCATIONS:
Overall Officials: Tsai-Wei Huang, PhD, Study Chair — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei County, Taiwan